CLINICAL TRIAL: NCT03211026
Title: Urinary Tract Infections in Kidney Transplant Recipients : an Observational Cohort
Brief Title: Urinary Tract Infections in Kidney Transplant Recipients
Acronym: URIKIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-A02081-50
Record Dates: First submitted 2017-06-23; First posted 2017-07-07 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Kidney Transplantation
Keywords: Urinary tract infection; Multidrug resistant bacteria; Candiduria; Epidemiology; Graft rejection; Solid organ transplantation
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to better estimate the prevalence of urinary tract infections (UTI) in kidney transplant (KIT) recipients, and especially multidrug resistant (MDR) bacteria. KIT recipients have a higher risk of UTI over the 6 first months following the transplantation. Urine culture was done in a city lab or at hospital. Current data on bacteriuria and candiduria lead mostly to hospital data that are incomplete..

DETAILED DESCRIPTION:
The risk of UTI after a kidney transplantation is higher than in the general population. MDR bacteria, such as extended spectrum betalactamase (ESBL)-producing enterobacteriaceae or MDR Pseumomoas aeruginosa are emerging threats due to antibiotic selective pressure. Epidemiological data are mostly data from hospital laboratories that do not show a complete overview of the current situation. In addition, the different centers which participated to this study received before the beginning of the study a protocol to avoid carbapenem use. The main objective of this study is to assess the prevalence of MDR bacteria in an adult population of KIT recipients. Through this study, the management of UTI in KIT recipients will be improved. Data on bacteria or yeasts responsible for UTI (identification, resistance profile), antibiotic use, patients' outcome, and graft outcome will be collected.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 year-old
* Kidney transplanted for less than 5 years
* First symptomatic episode of UTI with bacteria or yeast
* To have a health insurance

Exclusion criteria

* Asymptomatic bacteriuria or candiduria
* Protected people
* Pregnant women -> 2 bacteria in the urinalysis without external or internal urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2022-05-04 (Estimated); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of UTI due to MDR bacteria | Day 0 to 2 years
  Proportion of MDR bacteria compared to other bacteria found in urinalysis of symptomatic KIT patients

SECONDARY OUTCOMES:
Epidemiology of UTI in KIT recipients | Day 0 to 2 years
  Frequency of each bacteria or yeasts responsible for UTI
Risk factors for MDR UTI | Day 0 to 2 years
  Comparison of demographic and clinical characteristic of patients who develop an MDR versus a non-MDR UTI
Carbapenem use to treat UTI | Day 0 to 2 years
  Proportion of patients who received carbapenem for UTI treatment
Coherence between antibiotic protocol and treatment received to treat UTI | Day 0 to 2 years
  Proportion of patients who received carbapenem while responsible bacteria was susceptible to other antibiotics
UTI relapse frequency | Day 0 to 2 years
  Proportion of patients with at least one relaspe of UTI with the same bacteria
UTI recurrence frequency with a different micororganism | Day 0 to 2 years
  Proportion of patients with more than one UTI during the study period
Assessment of kidney function during the observation period | Day 0 to 2 years
  Difference between the initial kidney function (MDRD) and the final kidney function at the end of the observation period
Graft outcome | Day 0 to 2 years
  Number of patients needed a dialysis
Patients outcome | Day 0 to 2 years
  Number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Antoine THIERRY, PHD, Principal Investigator — Poitiers University Hospital; Blandine RAMMAERT, Study Director — Poitiers University Hospital
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No
No plan will be sharing with others researchers